CLINICAL TRIAL: NCT02693847
Title: Natural History of Liver Cirrhosis Diagnosed by Transient Elastography in HIV/HCV-coinfected Patients
Status: Completed | Type: Observational
Sponsor: Hospital Universitario de Valme (Other)
Collaborators: Hospital Universitario Virgen Macarena (Other); Complejo Hospitalario Universitario de Huelva (Other); Hospital de La Línea (Unknown); Hospital Universitario Reina Sofia de Cordoba (Other Government); Hospital Universitario Virgen de la Victoria (Other); Complejo Hospitalario de Jaén (Unknown); Hospital Universitario Puerto Real (Other)
Responsible Party: Principal Investigator, Nicolás Merchante, MD, PhD, Hospital Universitario de Valme
Other Study IDs: HEPAVIR-Cirrhosis Cohort
Record Dates: First submitted 2015-11-24; First posted 2016-02-29 (Estimated); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Liver Cirrhosis; Hepatocellular Carcinoma; HIV; HCV Coinfection
Keywords: HCV; HIV; Liver cirrhosis; Hepatocellular carcinoma; Liver transplant; Liver stiffness; Transient elastography
MeSH Terms: conditions — Liver Cirrhosis; Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples Without DNA — Serum samples are collected and immediately frozen for criopreservation
Oversight: Data Monitoring Committee: No

SUMMARY:
Prospective multicenter cohort recruiting consecutive patients from 7 hospitals in Andalusia, southern Spain, according to following criteria: 1) HIV infection, 2) Chronic active HCV infection, 3) Older than 18 years, 4) New diagnosis of liver cirrhosis on the basis of a liver stiffness above 14 kiloPascals, 5) No previous or concomitant decompensation of liver disease. Patients are prospectively followed-up according to a uniform protocol of care. Epidemiological, clinical and laboratory variables are periodically recorded. The primary outcomes are the emergence of a liver decompensation (including hepatocellular carcinoma), liver transplant or death. The predictors of these outcomes are analyzed.

ELIGIBILITY:
Inclusion Criteria:

* HIV Infection
* HCV chronic active infection (positive serum RNA HCV at inclusion)
* New diagnosis of cirrhosis on the basis of a liver stiffness equal or greater than 14 kiloPascals.
* No previous or concomitant decompensation of liver disease

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV/HCV-coinfected patients diagnosed of cirrhosis on the basis of a liver stiffness equal or greater than 14 kiloPascals
Sampling Method: Probability Sample
Enrollment: 446 (Actual)
Dates: Start 2006-02; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who developed a first liver decompensation of cirrhosis during follow-up | 3 years
  Episodes of liver decompensation will include those episodes of ascites, spontaneous bacterial peritonitis, portal hypertensive gastrointestinal bleeding, hepatorrenal syndrome, hepatic encephalopathy, hepatocellular carcinoma, non obstructive jaundice and acute on chronic liver failure. These episodes will be diagnosed according to standard definitions of clinical practice guidelines in the field (i.e. HCC diagnosis will be diagnosed according to AASLD criteria, spontaneous bacterial peritonitis and hepatorenal syndrome will be diagnosed following the EASL criteria, portal hypertensive gastrointestinal bleeding according Baveno VI consensus definition,…)

SECONDARY OUTCOMES:
Liver-related mortality | 3 Years
  Probability of liver-related death after enrollment
All cause mortality | 3 Years
  Probability of death of any cause

CONTACTS AND LOCATIONS:
Overall Officials: Nicolás Merchante, MD PhD, Principal Investigator — Andaluz Health Service
Locations (8):
- Spain (8):
  - Hospital de La Línea de la Concepción, La Línea de la Concepción, Cádiz
  - Hospital Universitario de Puerto Real, Puerto Real, Cádiz
  - Hospital Universitario Reina Sofía, Córdoba
  - Complejo Hospitalario de Huelva, Huelva
  - Complejo Hospitalario de Jaén, Jaén
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario de Valme, Seville
  - Hospital Universitario Virgen Macarena, Seville

REFERENCES:
- [Result] Merchante N, Rivero-Juarez A, Tellez F, Merino D, Jose Rios-Villegas M, Marquez-Solero M, Omar M, Macias J, Camacho A, Perez-Perez M, Gomez-Mateos J, Rivero A, Antonio Pineda J; Grupo Andaluz para el Estudio de las Hepatitis Viricas (HEPAVIR) de la Sociedad Andaluza de Enfermedades Infecciosas (SAEI). Liver stiffness predicts clinical outcome in human immunodeficiency virus/hepatitis C virus-coinfected patients with compensated liver cirrhosis. Hepatology. 2012 Jul;56(1):228-38. doi: 10.1002/hep.25616. Epub 2012 Jun 6. PMID 22278746
- [Result] Recio E, Macias J, Rivero-Juarez A, Tellez F, Merino D, Rios M, Marquez M, Omar M, Rivero A, Lorenzo S, Merchante N, Pineda JA. Liver stiffness correlates with Child-Pugh-Turcotte and MELD scores in HIV/hepatitis C virus-coinfected patients with cirrhosis. Liver Int. 2012 Jul;32(6):1031-2. doi: 10.1111/j.1478-3231.2012.02782.x. Epub 2012 Mar 9. No abstract available. PMID 22405076
- [Result] Pineda JA, Recio E, Camacho A, Macias J, Almodovar C, Gonzalez-Serrano M, Merino D, Tellez F, Rios MJ, Rivero A; Grupo Andaluz de Hepatitis Virica (HEPAVIR) de la Sociedad Andaluza de Enfermedades Infecciosas (SAEI). Liver stiffness as a predictor of esophageal varices requiring therapy in HIV/hepatitis C virus-coinfected patients with cirrhosis. J Acquir Immune Defic Syndr. 2009 Aug 1;51(4):445-9. doi: 10.1097/QAI.0b013e3181acb675. PMID 19487952
- [Result] Merchante N, Tellez F, Rivero-Juarez A, Rios-Villegas MJ, Merino D, Marquez-Solero M, Omar M, Recio E, Perez-Perez M, Camacho A, Macias-Dorado S, Macias J, Lorenzo-Moncada S, Rivero A, Pineda JA; Grupo Andaluz para el Estudio de las Hepatitis Viricas (HEPAVIR) de la Sociedad Andaluza de Enfermedades Infecciosas (SAEI). Progression of liver stiffness predicts clinical events in HIV/HCV-coinfected patients with compensated cirrhosis. BMC Infect Dis. 2015 Dec 7;15:557. doi: 10.1186/s12879-015-1291-3. PMID 26643257
- [Result] Merchante N, Rivero-Juarez A, Tellez F, Merino D, Rios-Villegas MJ, Ojeda-Burgos G, Omar M, Macias J, Rivero A, Perez-Perez M, Raffo M, Lopez-Montesinos I, Marquez-Solero M, Gomez-Vidal MA, Pineda JA; Grupo Andaluz para el Estudio de las Hepatitis Viricas (HEPAVIR) de la Sociedad Andaluza de Enfermedades Infecciosas (SAEI). Liver stiffness predicts variceal bleeding in HIV/HCV-coinfected patients with compensated cirrhosis. AIDS. 2017 Feb 20;31(4):493-500. doi: 10.1097/QAD.0000000000001358. PMID 27922855
- [Result] Merchante N, Aldamiz-Echevarria T, Garcia-Alvarez M, Rivero-Juarez A, Macias J, Miralles P, Jimenez-Sousa MA, Mancebo M, Perez-Latorre L, Pineda-Tenor D, Berenguer J, Resino S, Pineda JA. Bacterial translocation and clinical progression of HCV-related cirrhosis in HIV-infected patients. J Viral Hepat. 2018 Feb;25(2):180-186. doi: 10.1111/jvh.12769. Epub 2017 Sep 7. PMID 28783247
- [Result] Merchante N, Rivero-Juarez A, Tellez F, Merino D, Rios-Villegas MJ, Villalobos M, Omar M, Rincon P, Rivero A, Perez-Perez M, Raffo M, Lopez-Montesinos I, Palacios R, Gomez-Vidal MA, Macias J, Pineda JA; Members of the HEPAVIR-Cirrhosis Study Group. Sustained virological response to direct-acting antiviral regimens reduces the risk of hepatocellular carcinoma in HIV/HCV-coinfected patients with cirrhosis. J Antimicrob Chemother. 2018 Sep 1;73(9):2435-2443. doi: 10.1093/jac/dky234. PMID 29982683
- [Result] Merchante N, Saroli Palumbo C, Mazzola G, Pineda JA, Tellez F, Rivero-Juarez A, Rios-Villegas MJ, Maurice JB, Westbrook RH, Judge R, Guaraldi G, Schepis F, Perazzo H, Rockstroh J, Boesecke C, Klein MB, Cervo A, Ghali P, Wong P, Petta S, De Ledinghen V, Macias J, Sebastiani G. Prediction of Esophageal Varices by Liver Stiffness and Platelets in Persons With Human Immunodeficiency Virus Infection and Compensated Advanced Chronic Liver Disease. Clin Infect Dis. 2020 Dec 31;71(11):2810-2817. doi: 10.1093/cid/ciz1181. PMID 31813962